CLINICAL TRIAL: NCT05985304
Title: Clinical Trial to Investigate the Safety and Effectiveness of a Hydrophilic EMV Toric Lens RAO210T in the Correction of Aphakia and Post-operative Corneal Astigmatism
Brief Title: Clinical Trial of a Hydrophilic EMV Toric Lens RAO210T in the Correction of Aphakia and Corneal Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rayner Intraocular Lenses Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WR-2023-US-03
Record Dates: First submitted 2023-07-19; First posted 2023-08-14 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cataract; Corneal Astigmatism
Keywords: Toric Intraocular Lens
MeSH Terms: conditions — Cataract; Astigmatism | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Toric (test) group (Experimental): All subjects randomized to be implanted with the low cylinder (1.50 D) RayOne EMV Toric IOL (Model RAO210T)
  Interventions: Device: RayOne EMV Toric IOL; Procedure: Cataract Surgery
- Monofocal (control) group (Active Comparator): All subjects randomized to be implanted with the RAO600C Monofocal IOL
  Interventions: Device: RayOne Monofocal IOL; Procedure: Cataract Surgery

INTERVENTIONS:
Device: RayOne EMV Toric IOL — Implantation of intraocular lens.
  Other Names: Model RAO210T
  Arms: Toric (test) group
Device: RayOne Monofocal IOL — Implantation of intraocular lens.
  Other Names: RAO600C
  Arms: Monofocal (control) group
Procedure: Cataract Surgery — Removal of natural crystalline lens due to cataracts

SUMMARY:
The objectives of the clinical investigation are to determine the safety and performance of the RayOne EMV Toric (Model RAO210T) following unilateral implantation and approximately 6 months (120 to 180 days) of post-operative assessment, as a randomized comparison to aspheric monofocal control for low cylinder (1.50 D). This patient population with cataracts and low corneal cylinder (+1.00 to +1.50 D) will have the natural crystalline lens removed and replaced with an intraocular lens in the capsular bag.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, active controlled, masked (assessor and subject) pivotal investigation for unilateral implantation of low cylinder (1.50 D) toric IOL. It compares the Rayner RAO210T toric IOL to the Rayner RAO600C aspheric monofocal IOL. Subjects who sign the ICF are considered enrolled in the study. After signing the ICF, subjects will be screened for eligibility. Inclusion and Exclusion Criteria must be applied prior to subject randomization. Subjects who meet all protocol-specified eligibility criteria will be assigned to the randomized controlled study arms if the study eye's estimated IOL cylinder power using Barrett Toric Calculator is 1.50 D. Randomized subjects receive either the Rayner RAO210T Toric IOL (1.50 D low cylinder) or the Rayner RAO600C aspheric monofocal IOL in the study eye.

Up to 295 adult subjects will be enrolled (consented) assuming a 15% screen failure rate, then up to 250 subjects will be randomized, of which approximately 125 subjects will be randomized to receive low cylinder (1.50 D) RayOne EMV Toric (Model RAO210T) in one eye and approximately 125 subjects randomized to receive the RAO600C aspheric monofocal IOL in one eye, to complete 120-180 days follow-up for at least 100 subjects in each group.

All subjects who meet inclusion criteria will be assigned to the randomized controlled study arms to receive either the RAO210T toric IOL (1.50 D low cylinder) or the RAO600C aspheric monofocal IOL in the study eye according to a 1:1 ratio. Randomization will be stratified by site.

Up to 11 U.S. sites will be encouraged to enroll a minimum of 20 subjects. No site will enroll more than 25% of the subjects enrolled in the study.

If a subject has significant cataract in both eyes, it is recommended that cataract surgery is performed in one eye before the subject is enrolled in the study. Once a subject has been enrolled, it is recommended that the fellow eye does not undergo cataract surgery (except for a YAG capsulotomy) throughout the duration of the study. At screening, if both eyes qualify for the study, the eye to undergo cataract surgery and IOL implantation is the eye with worse pre-operative BCDVA. If pre-operative BCDVA is the same for each eye, the right eye will be the study eye.

Subjects will complete 6 study visits in approximately 9 months. Subject participation is calculated as the difference between the time of the pre-operative visit to completion of Visit 4 (120 to 180 days post-operative).

Standard clinical trial methods will be used to minimize bias, such as the use of site personnel performing manifest refraction and visual acuity assessments masked to subject treatment assignment, masking of subjects in the randomized controlled investigation evaluating low cylinder power, standardized test procedures, common Investigator training and common inclusion and exclusion criteria.

In order to minimize bias, measures will be taken to mask the site personnel performing post-operative manifest refraction and visual acuity assessments, as to the subject's treatment assignment until after the final database lock. Every attempt should be made to have the same masked site personnel perform the same masked post-operative assessments for an individual subject throughout the subject's study participation.

Subjects will be masked to their IOL assignment in the randomized controlled investigation evaluating low cylinder power. All material which may indicate the subjects' assignment, e.g., packaging, documents, etc., will be removed from any areas where subjects and/or masked site personnel may see them. Unmasked personnel will further be instructed to scrupulously avoid conversation and communication with masked personnel, subjects and all other persons regarding subjects' assignments, outcomes, clinical courses, and all other information potentially relevant to the study and its conduct.

Study Groups:

* Toric (test) group - all subjects randomized to be implanted with the low cylinder (1.50 D) RayOne EMV Toric IOL (Model RAO210T)
* Monofocal (control) group - all subjects randomized to be implanted with the RAO600C Monofocal IOL

Sample Size Determination:

Subjects will be enrolled with the goal of completing a total of 200 subjects through Visit 4 within the randomized groups, of whom 100 were implanted with the low cylinder RayOne EMV Toric IOL (Model RAO210T) and 100 were implanted with the RAO600C monofocal IOL.

Effectiveness For effectiveness, 100 subjects (eyes) randomized to the Toric (test) group (lowest cylinder power +1.50D) and 100 subjects (eyes) randomized to the Monofocal (control) group completing Visit 4 yields over 98% statistical power to reject H0e in favor of H1e and conclude the Toric IOL has statistically significantly lower mean residual manifest cylinder at Visit 4 compared to the Monofocal IOL, using a one-sided t-test with an alpha level of 0.025 and assuming a true mean difference of 0.4 D and a standard deviation of 0.7 D in both groups.

Safety For safety, ISO 11979-7 and ANSI Z80.30 specifies that a minimum of 100 subjects should complete a clinical evaluation of an IOL, where a parent IOL has been approved, to obtain appropriate specificity around adverse event and visual acuity rates.

Handling of Missing Data:

Missing data will be imputed for selected endpoints using the methods specified under the analysis descriptions for the endpoints. Where possible, multiple imputation will be used. Except where mentioned in Section 7, missing data will not be imputed.

Multiplicity Considerations:

The overall type I error rate for the toric effectiveness analyses will be controlled at 0.05. The study will be considered successful if all of the primary effectiveness and safety endpoints are met. Thus, no adjustments for multiplicity are necessary.

All primary effectiveness and primary safety endpoints as described below are required to achieve successful outcomes in order to demonstrate study success.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 22 years or older at the pre-operative visit who have cataract with best corrected distance visual acuity of 0.30 logMAR (20/40) or worse in at least one eye with or without a glare source present who are eligible for phacoemulsification cataract surgery
2. Subjects who are projected to have best corrected distance visual acuity 0.20 logMAR (20/30) or better after IOL implantation by potential acuity meter (PAM) or Investigator estimation
3. Clear intraocular media other than cataract
4. Contact lens wearers must demonstrate stability of biometry
5. Have the capability to understand and sign an IRB approved informed consent form and privacy authorization in accordance with local regulations
6. Female subjects must be 1-year postmenopausal, surgically sterilized, or, if of childbearing potential, have a negative urine pregnancy test at the Pre-operative Visit. Women of childbearing potential must use an acceptable form of contraception throughout the study.

   Acceptable methods include at least one of the following: intrauterine (intrauterine device), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.
7. Have Investigator selected IOL spherical equivalent power between +10.0 D to +25.0 D in 0.5 D steps and IOL cylinder power of +1.50 D
8. Have pre-existing corneal astigmatism of 1.00 D to 1.50 D as determined by keratometry
9. Dilated pupil size 5.5 mm or greater to allow visualization of the toric IOL axis markings post-operatively

Exclusion Criteria:

1. Previous intraocular, corneal, or retinal detachment surgery, including corneal transplant, LASIK / LASEK / PRK, SMILE, astigmatic keratotomy and limbal relaxing incisions in the planned operative eye.
2. Diagnosed degenerative visual disorders (e.g. macular degeneration, retinal detachment, proliferative diabetic retinopathy, or other retinal disorders) that are predicted to cause future acuity losses to a level of 0.20 logMAR (20/30) or worse
3. Significant anterior segment pathology that might increase intraoperative risk or compromise IOL stability (e.g. pseudoexfoliation syndrome, any iris pathology)
4. Subjects with conditions associated with increased risk of zonular rupture (that may affect post-operative centration or tilt of IOL) in the planned operative eye
5. Potentially occludable angle or ciliary body tumor, or other pathology that might increase risk to subject safety, based on gonioscopic observation
6. Subjects reasonably expected to require secondary ocular surgical intervention or laser treatment (other than YAG capsulotomy)
7. Subjects with clinically significant corneal pathology, potentially affecting corneal topography
8. Subjects with traumatic cataract in the planned operative eye
9. Participating in a concurrent drug or device clinical trial or who have participated in a drug or device trial within 30 days of the pre-operative visit
10. Subjects with any other serious ocular pathology (e.g. glaucoma, severe dry eye, history of intraocular inflammation, history of retinal surgery or retinal laser procedure) or underlying systemic medical condition (e.g., uncontrolled diabetes) or circumstance that, based on the Investigator's judgment, poses a concern for the subjects' safety or could confound the results of the study (History of cataract surgery with PC-IOL in one eye is allowed.)
11. Use of medications known to interfere with visual performance, pupil dilation, or iris structure within 30 days of the pre-operative visit, at the discretion of the Investigator
12. Pregnant or nursing females
13. Irregular astigmatism in the planned operative eye

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Packer, MD, Study Chair
Locations (9):
- United States (9):
  - Vold Vision, Fayetteville, Arkansas
  - ICON Eyecare, Grand Junction, Colorado
  - Vance Thompson Vision Alexandria, Alexandria, Minnesota
  - Moyes Eye Center, Kansas City, Missouri
  - Vance Thompson Vision North Dakota, West Fargo, North Dakota
  - Cleveland Eye Clinic, Avon, Ohio
  - Carolina Eyecare Physicians, Mt. Pleasant, South Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Parkhurst NuVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD will be made available to U.S. FDA for supporting premarket approval, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after device approval in the US
Access Criteria: To be determined by the study sponsor after device approval.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 274 enrolled subjects, 32 subjects were screen failures who did not meet the study-specific inclusion/exclusion criteria (32/274, 11.7%), five subjects were withdrawn before randomization (5/274, 1.7%)
Period: Overall Study
Arm/Group | Toric (Test) Group | Monofocal (Control) Group
Started | 118 | 120
Completed | 117 | 116
Not Completed | 1 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Subject was not implanted with the study device | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Toric (Test) Group | Monofocal (Control) Group | Total
Number analyzed (Participants) | 118 | 120 | 238
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 23 | 59
  >=65 years | 82 | 97 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (7.4) | 69.4 (7.0) | 68.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 70 | 136
  Male | 52 | 50 | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Black or African American | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 112 | 115 | 227
  Multiple | 0 | 2 | 2
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 115 | 116 | 231
Region of Enrollment [Number; unit: participants]
  United States | 118 | 120 | 238
Study Eye [Count of Participants; unit: Participants]
  Right Eye (OD) | 62 | 73 | 135
  Left Eye (OS) | 56 | 47 | 103
Axial Length [Mean (Standard Deviation); unit: mm] | 24.183 (1.118) | 24.120 (1.117) | 24.151 (1.116)
Anterior Chamber Depth [Mean (Standard Deviation); unit: mm] | 3.337 (0.401) | 3.247 (0.381) | 3.292 (0.393)
Uncorrected Distance Visual Acuity (UCDVA) [Mean (Standard Deviation); unit: logMAR] — Population: Subjects with a Uncorrected Distance Visual Acuity (UCDVA) measurement of 'Count Fingers' or 'Hand Motion' are excluded from logMAR summaries
  logMAR
    number analyzed (Participants) | 116 | 116 | 232
    (all) | 0.632 (0.407) | 0.556 (0.363) | 0.594 (0.387)
Best-corrected Distance Visual Acuity (BCDVA) Without Glare [Mean (Standard Deviation); unit: logMAR] | 0.183 (0.159) | 0.227 (0.236) | 0.205 (0.202)
Best-corrected Distance Visual Acuity (BCDVA) with Glare [Mean (Standard Deviation); unit: logMAR] — Population: Best-corrected Distance Visual Acuity (BCDVA) with Glare was only measured if BCDVA without Glare was better than 0.3 logMAR (20/40 Snellen).
  logMAR
    number analyzed (Participants) | 87 | 87 | 174
    (all) | 0.860 (0.569) | 0.866 (0.536) | 0.863 (0.551)
Keratometric Cylinder [Mean (Standard Deviation); unit: Diopter] | 1.206 (0.146) | 1.247 (0.136) | 1.227 (0.142)
Preoperative Keratometric Cylinder Subgroup [Count of Participants; unit: Participants]
  1.0 to <1.25 D | 76 | 63 | 139
  1.25 to 1.5 D | 42 | 57 | 99
Manifest Refraction Cylinder [Mean (Standard Deviation); unit: Diopter] | -1.121 (0.726) | -1.038 (0.592) | -1.079 (0.662)
Manifest Refraction Spherical Equivalent (MRSE) at 4m [Mean (Standard Deviation); unit: Diopter] | -1.4015 (2.9906) | -0.8896 (2.7307) | -1.1434 (2.8680)
Manifest Refraction Optical Infinity Spherical Equivalent (MROISE) [Mean (Standard Deviation); unit: Diopter] | -1.6472 (2.9851) | -1.1396 (2.7307) | -1.3913 (2.8649)
Target Postoperative (PO) Residual Astigmatism [Mean (Standard Deviation); unit: Diopter] — Population: One subject did not have a Barrett Toric Calculator entry
  Diopter
    number analyzed (Participants) | 117 | 120 | 237
    (all) | 0.183 (0.102) | 0.199 (0.127) | 0.191 (0.115)
Intraocular Lens (IOL) Power Spherical Equivalent (SE) [Mean (Standard Deviation); unit: Diopter] — Population: One subject did not have a Barrett Toric Calculator entry
  Diopter
    number analyzed (Participants) | 117 | 120 | 237
    (all) | 18.10 (3.29) | 18.55 (3.30) | 18.32 (3.29)
Target Residual Spherical Equivalent (SE) [Mean (Standard Deviation); unit: Diopter] — Population: One subject did not have a Barrett Toric Calculator entry
  Diopter
    number analyzed (Participants) | 117 | 120 | 237
    (all) | -0.012 (0.099) | -0.000 (0.120) | -0.006 (0.110)
LOCS III: Nuclear Color [Count of Participants; unit: Participants] — Nuclear Color (NC) was graded using the LOCS III photographic standards. Examiners selected one categorical grade (NC1-NC6) based on the reference images. Each category reflects increasing nuclear coloration/brunescence, with higher category numbers indicating greater severity. The study used categorical grades only. Results represent the number of participants in each NC category (Measure Type: Count of Participants; Unit: Participants). Population: One subject was randomized (Toric IOL) but not treated due to a Screen Failure upon re-screening
  Participants
    number analyzed (Participants) | 117 | 120 | 237
    NC1 | 14 | 14 | 28
    NC2 | 35 | 40 | 75
    NC3 | 50 | 50 | 100
    NC4 | 9 | 11 | 20
    NC5 | 8 | 2 | 10
    NC6 | 1 | 1 | 2
    NA | 0 | 2 | 2
LOCS III: Nuclear Opalescence [Count of Participants; unit: Participants] — Nuclear Opalescence (NO) was graded using the LOCS III photographic standards. Examiners selected one categorical grade (NO1-NO6) based on the reference images. Each category represents increasing nuclear opalescence (density/haziness), with higher category numbers indicating greater severity. The study used categorical grades only. Results represent the number of participants in each NO category (Measure Type: Count of Participants; Unit: Participants). Population: One subject was randomized (Toric IOL) but not treated due to a Screen Failure upon re-screening
  Participants
    number analyzed (Participants) | 117 | 120 | 237
    NO1 | 11 | 7 | 18
    NO2 | 31 | 38 | 69
    NO3 | 44 | 43 | 87
    NO4 | 6 | 7 | 13
    NO5 | 6 | 4 | 10
    NO6 | 1 | 0 | 1
    N/A | 18 | 21 | 39
LOCS III: Cortical Opacity [Count of Participants; unit: Participants] — Cortical Opacity (C) was graded using the LOCS III photographic standards. Examiners selected one categorical grade (C1-C5) based on cortical opacity patterns in the reference images. Each category reflects increasing cortical involvement, with higher numbers indicating greater severity.
  The study used categorical grades only. Results represent the number of participants in each C category (Measure Type: Count of Participants; Unit: Participants). Population: Although subjects qualified for the study, some layers of the lens did not present with cataract according to the LOCS scoring system and were marked as NA; therefore, this data is not available, and the number analyzed in row differs from the overall. Additionally, one subject was randomized (Toric IOL) but not treated due to a Screen Failure upon re-screening.
  Participants
    number analyzed (Participants) | 116 | 119 | 235
    C1 | 28 | 29 | 57
    C2 | 20 | 34 | 54
    C3 | 18 | 18 | 36
    C4 | 4 | 3 | 7
    C5 | 2 | 1 | 3
    NA | 44 | 34 | 78
LOCS III: Posterior Subcapsular [Count of Participants; unit: Participants] — Posterior Subcapsular Opacity (P) was graded using the LOCS III photographic standards. Examiners selected one categorical grade (P1-P5) based on the reference images. Each category reflects increasing posterior subcapsular opacity, with higher category numbers indicating greater severity. The study used categorical grades only. Results represent the number of participants in each P category (Measure Type: Count of Participants; Unit: Participants). Population: Although subjects qualified for the study, some layers of the lens did not present with cataract according to the LOCS scoring system and were marked as NA; therefore, this data is not available, and the number analyzed in row differs from the overall. Additionally, one subject was randomized (Toric IOL) but not treated due to a Screen Failure upon re-screening.
  Participants
    number analyzed (Participants) | 116 | 118 | 234
    P1 | 27 | 27 | 54
    P2 | 12 | 13 | 25
    P3 | 5 | 4 | 9
    P4 | 3 | 4 | 7
    P5 | 0 | 0 | 0
    NA | 69 | 70 | 139

OUTCOME MEASURES:

1. Primary Outcome: Mean Magnitude of Residual Manifest Cylinder
Description: Mean magnitude of residual manifest cylinder (as measured by manifest refractive cylinder).
Time Frame: 120 to 180 days post-operatively
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Toric (Test) Group | Monofocal (Control) Group
Number analyzed (Participants) | 117 | 116
Diopters | -0.368 (0.334) | -0.780 (0.532)

2. Primary Outcome: Adjusted Mean Difference Magnitude of Residual Manifest Cylinder
Description: The adjusted mean difference of residual manifest cylinder (as measured by manifest refractive cylinder) between Toric and Monofocal groups will be given together with a 95% confidence interval and associated one-sided p-value. This endpoint will be considered successful if the one-sided p-value ≤ 0.025.
Time Frame: 120 to 180 days post-operatively
Measure: Mean (95% Confidence Interval); unit: Diopters
Groups:
- Combined Toric and Control Groups: All subjects randomized to be implanted with the low cylinder (1.50 D) RayOne EMV Toric IOL (Model RAO210T) and RayOne Monofocal IOL (Model RAO600C)
  RayOne EMV Toric IOL: Implantation of intraocular lens. RayOne Monofocal IOL: Implantation of intraocular lens.
  Cataract Surgery: Removal of natural crystalline lens due to cataracts
Arm/Group | Combined Toric and Control Groups
Number analyzed (Participants) | 238
Diopters | -0.430 [-0.5441 to -0.3159]
Statistical Analysis 1: Comparison: Combined Toric and Control Groups; Test type: Superiority; p < 0.0001, ANCOVA

3. Primary Outcome: Axis Misalignment (Frequency and Percentage 10 Degrees)
Description: Frequency and percentage of RayOne EMV Toric (Model RAO210T) IOLs with IOL axis misalignment at Visit 4 (as determined by photographic method) less than 10 degrees.
Time Frame: 120 to 180 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Toric (Test) Group
Number analyzed (Participants) | 98
Participants | 92

4. Primary Outcome: Axis Misalignment (Frequency and Percentage 20 Degrees)
Description: Frequency and percentage of RayOne EMV Toric (Model RAO210T) IOLs with IOL axis misalignment at Visit 4 (as determined by photographic method) less than 20 degrees.
Time Frame: 120 to 180 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Toric (Test) Group
Number analyzed (Participants) | 98
Participants | 98

5. Primary Outcome: Stability of Toric IOL Axis Orientation (Frequency and Percentage)
Description: Stability of toric IOL axis orientation, expressed as frequency and percentage of RayOne EMV Toric (Model RAO210T) IOLs that rotate ≤ 5 degrees postoperatively between 30 to 60 days (Visit 3) and 120 to 180 days (Visit 4)
Time Frame: 30 to 60 days and 120 to 180 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Toric (Test) Group
Number analyzed (Participants) | 101
Participants | 100

6. Primary Outcome: Rates of IOL Adverse Events Per ISO 11979-7
Description: Rates of IOL adverse events through 120 to 180 days post-operatively (Visit 4) compared to the ISO Safety and Performance Endpoint (SPE) rates as described in ISO 11979-7.
  Rates of cumulative and persistent adverse events from ISO 11979-7 (2018) Table E.2 will be reported by treatment group (Toric test group, Monofocal control group) and AE type. Rates of adverse events will be compared to the SPE rate from Table E.2. The one-sided p-value from the exact binomial test of each hypothesis will also be provided for each adverse event. If none of these hypothesis test results are statistically significant, this endpoint will be considered successful for the toric IOL.
Time Frame: 120 to 180 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Toric (Test) Group | Monofocal (Control) Group
Number analyzed (Participants) | 117 | 116
Participants
  Cumulative - Cystoid macular edema | 2 | 1
  Cumulative - Hypopyon | 0 | 0
  Cumulative - Endophthalmitis | 0 | 0
  Cumulative - Lens dislocation from posterior chamber | 0 | 0
  Cumulative - Mechanical pupillary block | 0 | 0
  Cumulative - Retinal detachment | 0 | 0
  Cumulative - Secondary Surgical Intervention | 2 | 0
  Persistent - Cornea Stroma Edema | 0 | 0
  Persistent - Cystoid macular edema | 0 | 0
  Persistent - Iritis | 0 | 0
  Persistent - Increased IOP | 0 | 0

7. Primary Outcome: Rates of All Other Adverse Events Not Included in ISO 11979-7
Description: The eyes with at least one adverse event not included in the cumulative and persistent adverse events from ISO 11979-7 (2018) Table E.2 through 120 to 180 days post-operatively (Visit 4) will be presented by treatment group (Toric test group, Monofocal control group).
Time Frame: 120 to 180 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Toric (Test) Group | Monofocal (Control) Group
Number analyzed (Participants) | 117 | 116
Participants
  Cornea Stroma Edema | 6 | 5
  Increased IOP | 4 | 7
  IOL decentration/malposition resulting in secondary surgical intervention | 1 | 0
  Iris pigment epithelium loss | 1 | 0
  Progression or onset diabetic retinopathy | 1 | 0
  Retained lens material | 1 | 0
  Secondary Surgical Intervention - Wound burp (aqueous tap, or paracentesis) | 1 | 0
  Other - Posterior capsular opacification requiring YAG capsulotomy | 14 | 4
  Other - Posterior vitreous detachment | 7 | 11
  Other - Corneal edema | 7 | 7
  Other - Anterior chamber cells greater than Grade 2 at Visit 1 | 5 | 1
  Other - Corneal abrasion | 3 | 0
  Other - Epithelial defect | 2 | 1
  Other - Choroidal nevus | 1 | 1
  Other - Corneal dellen | 1 | 1
  Other - Dermatochalasis | 1 | 1
  Other - Epiretinal membrane | 2 | 0
  Other - Subconjunctival hemorrhage | 1 | 1
  Other - Worsening dry eye disease | 1 | 1
  Other - Central capsular wrinkle | 1 | 0
  Other - Chemosis | 1 | 0
  Other - Double vision secondary to neurological adjustment following cataract surgery | 1 | 0
  Other - Epithelial basement membrane dystrophy | 1 | 0
  Other - Intraretinal hemorrhage | 1 | 0
  Other - Photophobia | 1 | 0
  Other - Retinal pigment epithelial mottling | 1 | 0
  Other - Superficial punctate keratitis | 1 | 0
  Other - Trace punctate epithelial erosions | 1 | 0
  Other - Visually significant corneal edema resulting in BCDVA of 0.3 or worse | 1 | 0
  Other - Worsening punctate epithelial erosion | 1 | 0
  Other - Conjunctival injection | 0 | 2
  Other - Dry eye disease | 0 | 1
  Other - Iritis | 0 | 1
  Other - Keratoconjunctivitis Sicca, not specified as Sjogrens | 0 | 1
  Other - Retinal pigment epithelial changes | 0 | 1

8. Primary Outcome: Rates of Secondary Surgical Interventions for IOL Repositioning Due to IOL Misalignment
Description: The percentage of eyes implanted with the Toric test group IOL requiring a secondary surgical intervention for IOL repositioning due to IOL misalignment through 120 to 180 days post-operatively (Visit 4), as well as a two-sided 95% exact binomial confidence interval for the percentage, will be presented.
Time Frame: 120 to 180 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Toric (Test) Group
Number analyzed (Participants) | 117
Participants | 1

9. Primary Outcome: Rate of BCDVA of 0.30 logMAR or Better Compared to the ISO SPE Rates
Description: The percentage of eyes that achieve a BCDVA at 4 meters of 0.30 logMAR or better at 120 to 180 days post-operatively (Visit 4) will be presented by treatment group (Toric test group, Monofocal control group) for the Safety Set and Best Case Set. If neither of these hypothesis test results are statistically significant, this endpoint will be considered successful for the toric IOL.
Time Frame: 120 to 180 days post-operatively
Population: Toric subjects 01-003, 01-009, 01-026, 01-027, 01-030 and 05-009; and Monofocal subjects 07-031 and 08-036; are excluded from the PP Set due to Major Protocol Deviations.
  Per Protocol Monofocal subjects 02-006, 03-064, 05-012, 05-014 were excluded from the BCS due to significant pre-operative ocular pathology in the study eye. No Per Protocol Toric subjects were excluded from the BCS.
Measure: Count of Participants; unit: Participants
Arm/Group | Toric (Test) Group | Monofocal (Control) Group
Number analyzed (Participants) | 117 | 116
Participants
  Safety Set | 117 | 116
  Best Case Set: number analyzed (Participants) | 112 | 111
  Best Case Set | 112 | 111

10. Secondary Outcome: Residual Manifest Cylinder Stratified by Preoperative Keratometric Cylinder
Description: Residual manifest refractive cylinder by subgroups of 0.25 D preoperative keratometric cylinder at 120 to 180 days post-operatively
Time Frame: 120 to 180 days post-operatively
Measure: Mean (Standard Deviation); unit: Diopters
Groups:
- Toric (Test) Group With Low Preoperative Keratometric Cylinder: All subjects randomized to be implanted with the low cylinder (1.50 D) RayOne EMV Toric IOL (Model RAO210T) with low preoperative keratometric cylinder (1.0 to <1.25 D)
  RayOne EMV Toric IOL: Implantation of intraocular lens.
  Cataract Surgery: Removal of natural crystalline lens due to cataracts
- Monofocal (Control) Group With Low Preoperative Keratometric Cylinder: All subjects randomized to be implanted with the RAO600C Monofocal IOL with low preoperative keratometric cylinder (1.0 to <1.25 D)
  RayOne Monofocal IOL: Implantation of intraocular lens.
  Cataract Surgery: Removal of natural crystalline lens due to cataracts
- Toric (Test) Group With High Preoperative Keratometric Cylinder: All subjects randomized to be implanted with the low cylinder (1.50 D) RayOne EMV Toric IOL (Model RAO210T) with low preoperative keratometric cylinder (1.25 to 1.5 D)
  RayOne EMV Toric IOL: Implantation of intraocular lens.
  Cataract Surgery: Removal of natural crystalline lens due to cataracts
- Monofocal (Control) Group With High Preoperative Keratometric Cylinder: All subjects randomized to be implanted with the RAO600C Monofocal IOL with low preoperative keratometric cylinder (1.25 to 1.5 D)
  RayOne Monofocal IOL: Implantation of intraocular lens.
  Cataract Surgery: Removal of natural crystalline lens due to cataracts
Arm/Group | Toric (Test) Group With Low Preoperative Keratometric Cylinder | Monofocal (Control) Group With Low Preoperative Keratometric Cylinder | Toric (Test) Group With High Preoperative Keratometric Cylinder | Monofocal (Control) Group With High Preoperative Keratometric Cylinder
Number analyzed (Participants) | 75 | 62 | 42 | 54
Diopters | -0.413 (0.333) | -0.794 (0.535) | -0.286 (0.325) | -0.764 (0.533)

11. Secondary Outcome: Percent Change in Absolute Cylinder Stratified by Preoperative Keratometric Cylinder
Description: Percent reduction in absolute cylinder (as measured by residual manifest cylinder / preoperative keratometric cylinder), at 120 to 180 days post-operatively. Positive numbers represent an decrease in cylinder and negative numbers represent an increase in cylinder.
Time Frame: 120 to 180 days post-operatively
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Toric (Test) Group | Monofocal (Control) Group
Number analyzed (Participants) | 117 | 116
percent change | 68.59 (29.17) | 36.11 (45.69)

ADVERSE EVENTS:
Time Frame: 6 months
Description: All AEs that occurred during or after the Pre-operative Visit through completion of study participation were recorded on the subject's case report form. The case report form included a list of anticipated AEs.
Arm/Group | Toric (Test) Group | Monofocal (Control) Group
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/116
Serious Adverse Events (participants affected / at risk) | 1/117 | 0/116
Other Adverse Events (participants affected / at risk) | 49/117 | 40/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Toric (Test) Group (N=117) | Monofocal (Control) Group (N=116)
Secondary Surgical Intervention - Surgical removal of retained lens fragment (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toric (Test) Group (N=117) | Monofocal (Control) Group (N=116)
Cornea Stroma Edema (Eye disorders) | 6 (6) | 5 (5)
Posterior capsular opacification requiring YAG capsulotomy (Eye disorders) | 14 (14) | 4 (4)
Posterior vitreous detachment (Eye disorders) | 7 (7) | 11 (11)
Corneal edema (Eye disorders) | 7 (7) | 7 (7)
Increased IOP (Eye disorders) | 4 (4) | 7 (7)
Anterior chamber cells greater than Grade 2 at Visit 1 (Eye disorders) | 5 (5) | 1 (1)
Corneal abrasion (Eye disorders) | 3 (3) | 0 (0)
Cystoid macular edema (Eye disorders) | 2 (2) | 1 (1)
Epithelial defect (Eye disorders) | 2 (2) | 1 (1)
Epiretinal membrane (Eye disorders) | 2 (2) | 0 (0)
Choroidal nevus (Eye disorders) | 1 (1) | 1 (1)
Corneal dellen (Eye disorders) | 1 (1) | 1 (1)
Dermatochalasis (Eye disorders) | 1 (1) | 1 (1)
Subconjunctival hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Worsening dry eye disease (Eye disorders) | 1 (1) | 1 (1)
Conjunctival injection (Eye disorders) | 0 (0) | 2 (2)
Central capsular wrinkle (Eye disorders) | 1 (1) | 0 (0)
Chemosis (Eye disorders) | 1 (1) | 0 (0)
Double vision secondary to neurological adjustment following cataract surgery (Eye disorders) | 1 (1) | 0 (0)
Epithelial basement membrane dystrophy (Eye disorders) | 1 (1) | 0 (0)
IOL decentration/malposition resulting in secondary surgical intervention (Eye disorders) | 1 (1) | 0 (0)
IOL repositioning (existing IOL is surgically moved to another location or rotated) (Eye disorders) | 1 (1) | 0 (0)
Intraretinal hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Iris pigment epithelium loss (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Progression or onset diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Retained lens material (Eye disorders) | 1 (1) | 0 (0)
Retinal pigment epithelial mottling (Eye disorders) | 1 (1) | 0 (0)
Superficial punctate keratitis (Eye disorders) | 1 (1) | 0 (0)
Surgical removal of retained lens fragment (Eye disorders) | 1 (1) | 0 (0)
Trace punctate epithelial erosions (Eye disorders) | 1 (1) | 0 (0)
Visually significant corneal edema resulting in BCDVA of 0.3 or worse (Eye disorders) | 1 (1) | 0 (0)
Worsening punctate epithelial erosion (Eye disorders) | 1 (1) | 0 (0)
Wound burp (aqueous tap, or paracentesis) (Eye disorders) | 1 (1) | 0 (0)
Dry eye disease (Eye disorders) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 0 (0) | 1 (1)
Keratoconjunctivitis Sicca, not specified as Sjogrens (Eye disorders) | 0 (0) | 1 (1)
Retinal pigment epithelial changes (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05985304/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05985304/SAP_001.pdf